CLINICAL TRIAL: NCT05015751
Title: Assessment Of Flow In Cerebrospinal Fluid Shunts With A Wireless Thermal Anisotropy Measurement Device: Phase A
Brief Title: Assessment of CSF Shunt Flow With Thermal Measurements A
Status: Completed | Type: Observational
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-01
Record Dates: First submitted 2021-08-10; First posted 2021-08-20 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Hydrocephalus Patients: Hydrocephalus patients with an existing ventriculoperitoneal shunt and symptoms of a shunt malfunction.
  Interventions: Device: Thermal Anisotropy Measurement Device

INTERVENTIONS:
Device: Thermal Anisotropy Measurement Device — A wireless device for non-invasively assessing CSF shunt flow.
  Other Names: FlowSense

SUMMARY:
This study evaluates the performance of a non-invasive thermal measurement device for assessing CSF shunt flow. Patients with an existing implanted shunt and symptoms of shunt malfunction will be evaluated with the study device.

DETAILED DESCRIPTION:
Patients with an existing implanted ventriculoperitoneal (VP) shunt and who are experiencing shunt malfunction symptoms will be recruited by the clinical investigators at each investigational site in accordance with the inclusion and exclusion criteria. Assessment of shunt flow will be performed non-invasively with the study device; physician and clinical staff will be blinded to the device result. Standard-of-care assessment of shunt function will be performed and surgical intervention will occur based on the judgement of the treating neurosurgeon without the use of study device data. This trial will evaluate the ability of the study device to identify shunt malfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Existing ventriculoperitoneal CSF shunt
* At least one symptom of shunt malfunction as determined by the investigator, including seizure, fever, headache, vision problems, dizziness, disorientation, confusion, vomiting, lethargy, irritability, difficulty waking or staying awake, swelling along shunt tract, enlargement of head, loss of balance, gait disturbance, and loss of sensory or motor function
* Suspicion of shunt obstruction warrants the performance of a test for this condition in the investigator's judgement
* Region of intact skin overlying an unambiguously identifiable chronically indwelling ventricular shunt which crosses the clavicle and is appropriate in size for application of the study device
* Available for follow-up for up to fourteen days
* Signed informed consent by patient or a parent, legal guardian, health care agent, or legally authorized representative.
* Verbal assent by minors four years of age and older who are able to understand the study and communicate their decision

Exclusion Criteria:

* Presence of multiple shunts, or presence of more than one distal shunt catheter (regardless of function) crossing the clavicle ipsilateral to the shunt with suspected obstruction
* Use of the study device would interfere with standard patient care, or emergency surgery that cannot be delayed
* Presence of an interfering open wound or edema over any portion of the shunt
* Patient-reported history of adverse skin reactions to adhesives
* Investigator judges that the subject is likely to be lost to follow-up due to unavailability or clinical outcome being unobtainable
* Participation in the study will interfere with, or be detrimental to, administration of optimal health-care to the subject
* Prior enrollment in this study (multiple enrollments of the same patient are disallowed)
* Participation in any other investigational procedural, pharmaceutical, and/or device study that may influence the collection of valid data under this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hydrocephalus patients with an existing ventriculoperitoneal shunt and shunt malfunction symptoms
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandi Lam, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (4):
- United States (4):
  - UCSF Benioff Children's Hospital - Oakland, Oakland, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois

REFERENCES:
- [Derived] Limbrick DD Jr, Skoch J, Auguste K, Grant GA, Lam SK, Tate MC, Langer DJ, Roland JL, Alden TD, Charbel FT, Lober RM, Patten K, Kennedy E, Farless C, Himsworth S, Fasbender R, Lovell-Ewen L, Morales DM, Correia CF, Burton A, Koschnitzky JE, Webb RC, Zysk AM. A Multicenter Study of Noninvasive Wireless Assessment of Cerebrospinal Fluid Shunt Function in Hydrocephalus Patients. Neurosurgery. 2025 Dec 1;97(6):1397-1405. doi: 10.1227/neu.0000000000003569. Epub 2025 Jun 16. PMID 40522244

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrocephalus Patients
Started | 44
Completed | 40
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Hydrocephalus Patients
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 3
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 3
  Race: White | 26
  Race: More than one Race | 1
  Race: Other | 3
  Race: Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Study Device Sensitivity
Description: Study device sensitivity is calculated as TP / (TP + FN), where TP = true positive and FN = false negative.
Time Frame: 14-day follow-up period
Measure: Number; unit: percent
Arm/Group | Hydrocephalus Patients
Number analyzed (Participants) | 23
percent | 88

2. Primary Outcome: Study Device Specificity
Description: Study device specificity is calculated as TN / (TN + FP), where TN = true negative and FP = false positive.
Time Frame: 14-day follow-up period
Measure: Number; unit: percent
Arm/Group | Hydrocephalus Patients
Number analyzed (Participants) | 23
percent | 87

ADVERSE EVENTS:
Time Frame: 20 minutes
Description: Patients were evaluated for adverse events during the use of the study device and for a period of 20 minutes thereafter.
Arm/Group | Hydrocephalus Patients
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT05015751/Prot_SAP_000.pdf